CLINICAL TRIAL: NCT02655796
Title: Evaluation of Screening Accuracy of a Device for Fall Risk Assessment in the Elderly: a Cross-sectional Study With a Futility Design
Brief Title: A Device for Screening of Fall Risk in the Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: OAK
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-02

CONDITIONS: Postural Imbalance; Gait, Unsteady
Keywords: Accidental Falls; Risk Assessment; Frail Elderly
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moderate/High Risk (Experimental): Participants assessed as moderate/high risk of falling according to the CDC Algorithm for Fall Risk Assessment
  Interventions: Device: OAK
- Low Risk (Experimental): Participants assessed as low risk of falling according to the CDC Algorithm for Fall Risk Assessment
  Interventions: Device: OAK

INTERVENTIONS:
Device: OAK — The OAK device evaluates the fall risk through exercises assessing mobility, equilibrium and postural reaction.

SUMMARY:
This study evaluates the screening accuracy of a device (OAK) in assessing fall risk in the elderly, compared to the assessment provided by the Algorithm for Fall Risk Assessment of the Centers for Disease Control and Prevention (CDC).

The OAK device is a technologic system, based on virtual reality. It allows to quickly perform a fall risk assessment integrating clinical indexes of the Brief-BESTest (The Balance Evaluation System Test), and kinematic and posturgraphic indexes. The participants interact with the OAK device through simple exercises, then the device provides an assessment of their functional mobility, equilibrium and postural reactions.

DETAILED DESCRIPTION:
Falls are a serious problem among the elderly. Most falls do not cause death, but 20%-30% of falls result in serious injuries representing a significant source of morbidity and mortality. Good evidence shows that many falls can be prevented. Thus, identifying people with risk of falling is crucial. The aim of this study is the evaluation of the screening accuracy of a device (OAK) in assessing fall risk in the elderly.

Participants are recruited at IRCCS Galeazzi Orthopedic Hospital in Milan, among outpatients and healthy volunteers. A brief questionnaire is administered in order to collect data relevant to the CDC Algorithm for Fall Risk Assessment. Then, participants are assessed through the OAK device. The OAK assessment is evaluated in terms of performance, accuracy (in comparison to the CDC Algorithm for Fall Risk Assessment) and safety.

ELIGIBILITY:
Inclusion Criteria:

* Able to walk without walking aids.
* Signed informed consent.

Exclusion Criteria:

* Neurological, musculoskeletal and orthopaedic disorders limiting mobility function and equilibrium. Psychiatric disorders. Any other medical condition limiting mobility function, as diabetes, obesity, serious ocular disorders (e.g. glaucoma), vestibular disorders (e.g. labyrinthitis) and proprioceptive disorders (e.g. ataxia).
* Pacemaker.
* Surgical interventions for orthopaedic disorders (e.g. knee or hip prosthesis) during the previous 6 months.
* Drug intake altering coordination and equilibrium (e.g. anti-epileptic, sedative-hypnotic drugs).
* Pregnancy.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 184 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
OAK failures in the fall risk assessment | Baseline
  Proportion of participants for which the OAK device is not able to provide a fall risk assessment
OAK sensitivity in the fall risk assessment | Baseline
  Proportion of participants assessed by the OAK device as moderate/high risk of falling among those at moderate/high risk according to the CDC Algorithm for Fall Risk Assessment

SECONDARY OUTCOMES:
Adverse events | Baseline
  Adverse events occurring during the assessment
Serious adverse events | Baseline
  Serious adverse events occurring during the assessment
Rate of falls | During the previous 6 months
  Number of falls during the prevoius 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Banfi, MD, Principal Investigator — banfi.giuseppe@fondazionesanraffaele.it
Locations (1):
- IRCCS Galeazzi Orthopedic Hospital, Milan, Italy

REFERENCES:
- [Derived] Castellini G, Gianola S, Stucovitz E, Tramacere I, Banfi G, Moja L. Diagnostic test accuracy of an automated device as a screening tool for fall risk assessment in community-residing elderly: A STARD compliant study. Medicine (Baltimore). 2019 Sep;98(39):e17105. doi: 10.1097/MD.0000000000017105. PMID 31574809